CLINICAL TRIAL: NCT03483766
Title: Individualized Robotic Functional Rehabilitation for Spinal Cord Injury
Brief Title: Robotic Rehabilitation for Spinal Cord Injury
Acronym: SCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: UW 17-307
Record Dates: First submitted 2018-03-20; First posted 2018-03-30 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2019-09

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: This study will apply spinal cord resting-state fMRI and DTI to patients with cervical spinal cord injury. Findings with fMRI/DTI will compare to clinical hand function evaluation by using American Spinal Injury Association (ASIA) with full ASIA sensory and motor examinations (International standards for neurological classification of spinal cord injury (ISNCSCI)). After baseline spinal cord MRI scan, those patients will receive 3 months muscle strength enhancement as pre-rehabilitation. Then, we will design robotic hand rehabilitation programme for each individuals. All participants will receive robotic rehabilitation for 1 year. After then, a follow-up spinal cord MRI scan and clinical assessment will evaluate the results of this project.
Who Masked: Investigator
Masking Description: Patients with tetraplegia under the care of our department will be recruited. Spinal cord resting-state fMRI and DTI, surface EMG tests from different muscles from arm will be detected to define 5 most possible suitable candidates for this project.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline before robotic functional rehabilitation (No Intervention): Baseline spinal cord MRI scan
- post rehabilitation (Experimental): Those patients will receive 3 months muscle strength enhancement as pre-rehabilitation. Then, we will design robotic hand rehabilitation programme for each individuals. All participants will receive robotic rehabilitation for 1 year. After then, a follow-up spinal cord MRI scan and clinical assessment will evaluate the results of this project.
  Interventions: Device: Robotic Functional Rehabilitation system

INTERVENTIONS:
Device: Robotic Functional Rehabilitation system — The tailored-made EMG driven soft-robotic hand prosthesis for tetraplegia individuals may help to preserve the residual function and to enhance the functional recovery.
  Arms: post rehabilitation

SUMMARY:
Individuals with spinal cord injury (SCI) have significant functional loss and poor quality of life. Individuals with cervical SCI are suffering much worse sickness within the SCI population. Tetraplegia resulting from cervical SCI bring a formidable emotional, physical, and financial burden in our society. Hand function is especially important to people with tetraplegia. Hand function is associated with independence in many activities, and impairments in upper extremity function can compound difficulties in many other areas, such as bowel and bladder management. Thus, it is not surprising that restoring hand function was found to be a priority for individuals with tetraplegia.

Nowadays, magnetic resonance imaging (MRI) plays an essential role in the diagnosis of SCI and helps to monitor disease progression and efficacy of therapies. Advanced MRI techniques, such as diffusion tensor imaging (DTI) and functional MRI (fMRI), have shown the potential to improve the understanding of human spinal cord in healthy and pathological condition, and serve as imaging biomarkers to characterize damage degree, monitor the response to treatment, and predict the outcome of intervention. Meanwhile, multi-channel EMG (Electromyography) recordings can provide a mapping of neuromuscular activities from an electrode-array.

The application of robotics in upper extremity function restoration of SCI patients has been started to help SCI patients to recovery upper extremity function. Combined DTI and fMRI to monitor the recovery of upper extremity function of SCI patients, this project will provide a tailored-made EMG driven soft-robotic hand prosthesis for tetraplegia individuals. We will provide the individuals with neuromuscular rehabilitation to preserve the residual function and to enhance the functional recovery. The eventual goal is to further design a useful robotic hand for regaining partial daily function to improve the quality of life for those individuals with tetraplegia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with tetraplegia under the care of Department of Orthopaedics and Traumatology, LKS Faculty of Medicine, The University of Hong Kong in Queen Mary Hospital.

Exclusion Criteria:

* Subjects with any neurological abnormality in brain, intellectual disability or other communication difficulty, subjects with pacemaker or metal implants, subjects with claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Spinal cord neuroimage | Changes between baseline on enrollment and 12 months follow-up
  Advanced MRI techniques, such as diffusion tensor imaging (DTI) and functional MRI (fMRI)

CONTACTS AND LOCATIONS:
Locations (1):
- The university of Hong Kong, Hong Kong, Hong Kong